CLINICAL TRIAL: NCT03452592
Title: Multicenter, Randomized and OpenⅡb Clinical Trials to Evaluate the Efficacy and Safety of Alflutinib in Locally Advanced or Metastatic Non-Small Cell Lung Cancer Patients Harbouring T790M Mutation
Brief Title: Efficacy and Safety of Alflutinib in Locally Advanced or Metastatic Non-Small Cell Lung Cancer Patients With T790M
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Indications have been approved for marketing
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180208
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Advanced NSCLC Patients With T790M
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The way patients take Alflutinib (Experimental): patients take Alflutinib orally once per day at dose of 80mg or160mg
  Interventions: Drug: Alflutinib

INTERVENTIONS:
Drug: Alflutinib — Patients take Alflutinib orally once per day at dose of 80 mg or 160 mg

SUMMARY:
This study is conducted to evaluate the efficacy and safety of Alflutinib in locally advanced or metastatic non-small cell lung cancer patients harbouring T790M mutation

DETAILED DESCRIPTION:
This is a multicenter, randomized and open Ⅱb phase study assessing the efficacy and safety of Alflutinib at doses of 80 mg orally /once daily and 160 mg orally /once daily in patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) harboring acquired T790M mutation after EGFR-TKI treatment or primary T790M mutation.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female, aged at least 18 years.
* 2.Histologically or cytologically confirmed, and locally advanced or metastatic NSCLC, who are not suitable for surgery /radiotherapy.
* 3.Patients who have disease progression after continuous previous treatment of 1st/2nd-generation EGFR TKIs (evaluation according to imaging evidence, judged by research center) will be recruited and primary T790M mutation patients are allowed to have received no EGFR-targeting therapy before detection.
* 4.The tissue/cell specimen collected from patients who have received the recent treatment (either TKI or chemotherapy) progression should be confirmed to T790M positive mutation by the detection of central laboratory, while no specimen collection requirements for the primary T790M mutation patients.
* 5. ECOG performance status of 0 to 2. Life expectancy of at least 12 weeks.
* 6. At least one measurable lesion by CT or MRI. The measureable lesion should receive no local treatments, such as, radiotherapy. If the lesions located at the regions which were previously treated are confirmed to progress, they can be chosen as lesion according to RECIST Version 1.1.
* 7. Organ function must meet the following requirements (patients should receive no blood transfusion, blood product, hematopoietic stimulating factors, and albumin)：

  * Absolute neutrophil count >= 1.5 x 109/L, Platelet count >= 75 x109/L, Haemoglobin >= 90 g/L;
  * Alanine aminotransferase/Aspartate aminotransferase <= 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or <= 5 times in the presence of liver metastases;
  * Total bilirubin <= 1.5 times ULN if no liver metastases or <= 3 times ULN in the presence of liver metastases;
  * Creatinine <=1.5 times ULN concurrent with creatinine clearance >= 50 ml/min (measured or calculated by Cockcroft and Gault equation);
* 8. Females who have fertility potential before menopause should have a pregnancy test in the time period of 7 days prior to start of dosing, should not be breast feeding and must have a negative pregnancy test (blood test or urinalysis) prior to start of dosing; all enrolled patients should take the barrier contraceptive methods during the therapy and three months after therapy
* 9. Patients are volunteered to enroll and sign a written informed consent form, and they can follow the therapeutic schedule and visit plan.

Exclusion Criteria:

* 1. Previous treatment as follows: Patients received any cytotoxic chemotherapy or immunotherapy (such as, PD-1 antibody, PD-L1antibody) from a previous treatment regimen or clinical study within 21 days prior to study entry; The time from stopping taking any target cancer drug of a previous treatment to study entry is less than its 5x half-life (such as, the time for erlotinib is less than 8 days, the time for gefinitib is less than 10 days, the time for icotinib is less than 2 days, the time for afatinib is less than 8 days ); The time from stopping taking any studied drug or anti-cancer drug of a previous treatment to study entry is less than its 5x half-life; Patients performed on major surgery within 4 weeks prior to study entry (excluding from and vascular passage-rebuilt surgery and biopsy operation); Patients performed on more than 30% of bone marrow radiotherapy or large area irradiation
* 2. Patients previously treated by 3nd-generation EGFR-TKI , analogous drug (such as Osimertinib (Tagrisso®, AZD9291), Rociletinib (CO-1686), Olmutinib (Olita®,HM61713), ASP8273, EGF816, HS-1029, and avitinib), or their bulk drugs and generic drug。
* 3. Patients were taking and could not stop the drugs within 2 weeks prior to study entry. The drugs are as following:

  * Potent inhibitors or inducers of CYP3A4;
  * Traditional Chinese medicine and preparations whose therapeutic goal is anti-tumors；Antitumor adjuvant therapy of Traditional Chinese medicine and preparations; Drugs with antitumor activity for patients judged by investigator.
* 4. Unrecovered toxic reaction due to former therapy existed, with over 1 grade of CTCAE (except alopecia) or 2 grade if ever applied DDP curing related neuropathy.
* 5. Spinal compression, or brain metastasis exhibiting symptoms but untreated (except those exhibit no symptom with stable condition and do not apply corticosteroids for 4 weeks before the trail initiating)
* 6. Any evidence showing severe or inadequate controlled systemic disease. For example patients with inadequate controlled hypertension considered not suitable for the trail or would affect the compliance towards the protocol, with active hemorrhagic tendency, with active infection such as HBV (HBV-DNA≥1000cps/ml), with HCV, with HIV et al (except for HBV carrier those the researcher considered meet the criterion).
* 7. Any condition affecting the drug taking, or significantly affecting the absorption or the pharmacokinetic parameters, include any kind of uncontrollable nausea or vomit, chronic gastroenteropathy, disability in swallowing, and history of gastrointestinal resection or surgery.
* 8. Any condition meet the following cardiac standard: ECG show a QTc>470 msec under resting state (Repeat in 48 hours when a first abnormal discovered, take mean of the two measurements). All kinds of abnormal in cardiac rhythm, conduction and resting ECG profile with clinical significance, for example complete left bundle branch block, 2 or 3 grade of conduction block and a PR interval>250 msec. Any possible factors increasing the risk of QTc extending or leading to arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, any first degree relative suffered from long QT syndrome or undertook unexplained sudden death before 40 years old, or taking any drug leading to a longer QTc.
* 9. Echocardiographic examination: LVEF<50%
* 10. Any history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonia require steroid therapy or active interstitial lung disease with clinical evidence during recruiting.
* 11. Lung functional examination: FEV1/FVC<70%, and FEV1<30%, or (DLCO%) < 40%.
* 12.Patients with acute onset or ongoing, pulmonary symptoms and interstitial lung disease that the researchers considered not suitable for trail.
* 13. Patients with other factors the researchers considered not suitable for the trail (for example, patients those who not willing to follow the procedure, limitation or requirements, who once experienced bone marrow allotransplantation, who have other kinds of malignant tumor coexisted or who showed allergic to the active ingredients or inactive adjuvant of the investigational drug, as well as drugs with similar chemical structure or in the same class).
* 14. Confirmed mutation of EGFR 20 exon insertion at anytime after the first diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Objective response rate of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks
  Evaluation of the objective response rate of Alflutinib in locally advanced or metastatic non-small cell lung cancer patients harbouring acquired T790M mutation by prior therapy with an EGFR-TKI or primary T790M mutation assessed by RECIST 1.1

SECONDARY OUTCOMES:
Progression free disease of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival
Overall survival of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks
  Evaluation of the overall survival of Alflutinib in locally advanced or metastatic non-small cell lung cancer patients harbouring acquired T790M mutation by prior therapy with an EGFR-TKI or primary T790M mutation assessed by RECIST 1.1
Duration of response of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks
  Evaluation of the duration of response of Alflutinib in locally advanced or metastatic non-small cell lung cancer patients harbouring acquired T790M mutation by prior therapy with an EGFR-TKI or primary T790M mutation assessed by RECIST 1.1
Disease control rate of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate disease control rate
Clinical benefit of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks
  Clinical benefit rate was calculated by adding up complete remission, partial remission and stabilization of disease assessed by RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- cancer hospital Chinese academy of medical sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Hu X, Zhang S, Lv D, Wu L, Yu Q, Zhang Y, Liu L, Wang X, Cheng Y, Ma Z, Niu H, Wang D, Feng J, Huang C, Liu C, Zhao H, Li J, Zhang X, Jiang Y, Gu C. Efficacy, safety, and genetic analysis of furmonertinib (AST2818) in patients with EGFR T790M mutated non-small-cell lung cancer: a phase 2b, multicentre, single-arm, open-label study. Lancet Respir Med. 2021 Aug;9(8):829-839. doi: 10.1016/S2213-2600(20)30455-0. Epub 2021 Mar 26. PMID 33780662